CLINICAL TRIAL: NCT03517787
Title: The Effect of Functional Electrical Stimulation and Therapeutic Exercise on Functional Properties of Skeletal Muscles, Sitting Postural Stability and Quality of Life in Traumatic Spinal Cord Injury Patients
Brief Title: The Effect of FES and Therapeutic Exercise on SCI Patients Skeletal Muscles, Sitting Balance, Posture and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Collaborators: University of Tartu (Other)
Responsible Party: Principal Investigator, Margot Bergmann, Junior research fellow of Physical Therapy, Tartu University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Spinaal
Record Dates: First submitted 2018-04-10; First posted 2018-05-07 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FES+TE (Experimental): Participants receiving Functional electrical stimulation (FES) combined with therapeutic exercise (TE)
  Interventions: Other: FES+TE
- TE (Active Comparator): Participants receiving only therapeutic exercise
  Interventions: Other: TE
- REF-FES+TE (Other): Healthy adults (reference group REF) that participate only in 1 session and receive FES and therapeutic exercise
  Interventions: Other: REF-FES+TE
- REF-TE (Other): Healthy adults that participate only in 1 session and receive only therapeutic exercise
  Interventions: Other: REF-TE

INTERVENTIONS:
Other: FES+TE — Group receive FES+therapeutic exercise during 6 weeks (twice a week). Altogether 8 exercises are conducted, each done 3 sets and 12 repetitions during first three weeks and 4 sets during last three weeks of intervention).
  Arms: FES+TE
Other: TE — Group perform only therapeutic exercise. Exercises are the same between all 4 groups.
  Arms: TE
Other: REF-FES+TE — Group perform FES+TE, but only participate in 1 session to collect reference data.
  Arms: REF-FES+TE
Other: REF-TE — Group perform only therapeutic exercise, but only participate in 1 session to collect reference data.
  Arms: REF-TE

SUMMARY:
Aim of the current study is to evaluate the effect functional electrical stimulation and therapeutic exercise on traumatic spinal cord injured participants'skeletal muscle characteristics, sitting balance, lung function and quality of life.

ELIGIBILITY:
Chronic spinal cord injury (12 months post injury) Injury in cervical region resulting in tetraparesis Able to sit on a custom made chair without support Does not have any contraindications for functional electrical stimulation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of median power frequency (MPF) and amplitude (A) | Change from baseline measure at 6 weeks
  Change of MPF and A is measured after first therapy to assess the baseline values and then after 6 weeks of therapy to assess the effectiveness of intervention.

SECONDARY OUTCOMES:
Change of muscle tone | Change from baseline measure at 6 weeks
  Muscle oscillation frequency (MOF) is measured to assess muscle tone. Change of MOF is measured after first therapy to assess the baseline values and then after 6 weeks of therapy to assess the effectiveness of intervention.

OTHER OUTCOMES:
Change of sitting balance | Change from baseline measure at 6 weeks
  Sitting balance is measured using Tekscan Conformat pressure mat. Static sitting balance is measured at a custom made stool, hands are placed on participants thighs. For dynamic sitting balance, participants are asked to move their center of pressure to 4 different directions. Distance is measured.
Health Related Quality of life | Change from baseline measure at 6 weeks
  RAND-36 questionnaire is used to measure health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Doris Vahtrik, Principal Investigator — University of Tartu
Locations (1):
- University of Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided